CLINICAL TRIAL: NCT03371251
Title: A Randomized Double-Blind Phase 1b/2 Combined Staggered Multiple Dose Escalation Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care
Brief Title: Study of BOS161721 in Systemic Lupus Erythematosus (SLE) Patients on a Background of Limited Standard of Care
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOS161721-02
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Adults; BOS161721; standard of care; moderately to severely active Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b: BOS161721 20, 60, 120 mg (Experimental): Participants will be randomized to receive a 20 milligram (mg), 60 mg, or 120 mg subcutaneous (SC) dose of BOS161721. Participants may receive a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
  Interventions: Drug: BOS161721
- Phase 1b: Placebo 20, 60, 120 mg (Placebo Comparator): Participants will be randomized to receive a 20 mg, 60 mg, or 120 mg SC dose of placebo. Participants may receive a total of 7 SC monthly doses of placebo on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
  Interventions: Drug: Placebo
- Phase 2: BOS161721 (Experimental): Participants will be randomized to receive a 120 mg SC dose of BOS161721 (as determined from Phase 1b of the study). Participants may receive a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
  Interventions: Drug: BOS161721
- Phase 2: Placebo (Placebo Comparator): Participants will be randomized to receive a 120 mg SC dose of placebo (as determined from Phase 1b of the study). Participants may receive a total of 7 SC monthly doses of placebo on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOS161721 — SC administration
  Arms: Phase 1b: BOS161721 20, 60, 120 mg; Phase 2: BOS161721
Drug: Placebo — SC administration
  Arms: Phase 1b: Placebo 20, 60, 120 mg; Phase 2: Placebo

SUMMARY:
This study will be conducted to assess the safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20 milligrams [mg], 60 mg, and 120 mg) administered subcutaneously in adult participants with moderately to severely active Systemic Lupus Erythematosus (SLE) on limited background standard of care treatment, in order to estimate the optimal dose.

BOS161721 at the chosen dose will be compared to placebo for response on the SLE Responder Index 4, with sustained reduction of oral corticosteroids, in the same participant population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 70 years, inclusive
* Participants must be mentally capable of giving consent and there must be evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study
* Participants must have Systemic Lupus Erythematosus (SLE) as defined by meeting 4 of the Systemic Lupus International Collaborating Clinics classification criteria for SLE (with at least 1 clinical and 1 immunologic criterion OR Lupus nephritis as the sole clinical criterion in the presence of anti-nuclear antibodies (ANA) or anti-double stranded deoxyribonucleic acid (dsDNA) antibodies), either sequentially or simultaneously
* At screening, participants must have at least 1 of the following:

  1. Elevated ANA ≥ 1:80 via immunofluorescent assay at the central laboratory
  2. Positive anti-dsDNA or anti-Smith (anti-Sm) above the normal level as determined by the central laboratory
* At screening, the total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score must be ≥ 8, including points from at least 1 of the following clinical components:

  a. Arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, and vasculitis Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.
* A clinical SLEDAI-2K score of ≥ 6 at screening at Day 0. Clinical SLEDAI-2K score is defined as follows:

  1. Contains points from arthritis, rash, myositis, mucosal ulcers, pleurisy, pericarditis, or vasculitis
  2. Excludes parameters which require central laboratory results: hematuria, pyuria, urinary casts, proteinuria, positive anti-dsDNA, decreased complement, thrombocytopenia, and leukopenia Note: Points from lupus headache and organic brain syndrome will also be excluded from qualifying total and clinical SLEDAI-2K scores at screening and Day 0.
* Participants must have at least 1 qualifying A or 2Bs from the following manifestations of SLE, as defined by the British Isles Lupus Assessment Group (BILAG) criteria as modified for use in this study, which must be confirmed by the central data reviewer:

  1. BILAG A or B score in the mucocutaneous body system. If a BILAG B score is due to BILAG number 6, mild skin eruption, the CLASI activity score including erythema and scale/hypertrophy must be ≥ 3 excluding points from mucosal ulcers and alopecia.
  2. BILAG A or B score in the musculoskeletal body system due to active polyarthritis Note: Hips, shoulders, back, neck, and temporomandibular joints do not count towards the total number of joints with active synovitis.

If only one "B" and no "A" score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 "B" must be present in at least 1 other body system for a total of 2 "B" BILAG body system scores.

- Participants must be currently receiving at least 1 of the following:

1. Administration for a minimum of 12 weeks, and a stable dose for at least 56 days (8 weeks prior to Day 0) of the following permitted steroid sparing agents: azathioprine (AZA), mycophenolate mofetil or mycophenolic acid, chloroquine, hydroxychloroquine, or methotrexate
2. If AZA, myocophenolate mofetil, mycophenolic acid, hydroxychloroquine, or MTX were discontinued prior to screening, the washout period must be ≥ 12 weeks.
3. Corticosteroids (CSs) (prednisone or prednisone-equivalent) at a stable dose of up to 30 mg/day for at least 6 weeks prior to Day 0

i. For participants whose only SLE treatment is CSs, the stable CS dose must be ≥ 10 mg/day for at least 6 weeks prior to Day 0 and no more than 30 mg/day at the time of randomization.

ii. Topical steroids may be used, but the dose must be stable for at least 6 weeks prior to Day 0. PRN topical steroids are not permitted.

* Women of childbearing potential (WOCBP):

  1. Must have a negative serum pregnancy test at screening. Urine pregnancy test must be negative prior to first dose
  2. Must not be breastfeeding
  3. Must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 52 weeks
* Participants must demonstrate willingness and ability to comply with the scheduled study visits, treatment plans, laboratory tests, and other procedures

Exclusion Criteria:

Participants presenting with any of the following will not be included in this study:

* Drug-induced SLE, rather than "idiopathic" SLE
* Other systemic autoimmune disease (eg, erosive arthritis, rheumatoid arthritis [RA], multiple sclerosis [MS], systemic sclerosis, or vasculitis not related to SLE). RA-Lupus overlap (Rupus), and secondary Sjogren syndrome are allowed.
* Any major surgery within 6 weeks of study drug administration (Day 0) or any elective surgery planned during the course of the study
* Any history or risk for tuberculosis (TB), specifically those with:

  1. Current clinical, radiographic, or laboratory evidence of active TB
  2. History of active TB
  3. Latent TB defined as positive QuantiFERON-TB Gold In Tube or other diagnostic test in the absence of clinical manifestations. Latent TB is not excluded if the participant has documented completion of adequate course of prophylactic treatment with regimen recommended by local health authority guideline, or the participant has started treatment with isoniazid, or other regimen recommended by local health authority guidelines for at least 1 month before Day 0 and continues to receive the prophylactic treatment during study until the treatment course is completed
* Active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria, with the exception of mononeuritis multiplex and polyneuropathy, which are allowed
* Severe proliferative lupus nephritis (World Health Organization Class III, IV), which requires or may require induction treatment with cytotoxic agents or high dose CSs
* Concomitant illness that, in the opinion of the investigator or the Sponsor or their designee, is likely to require additional systemic glucocorticosteroid therapy during the study, (eg, asthma), is exclusionary. However, treatment for asthma with inhalational CSs therapy is allowed.
* Use or planned use of concomitant medication outside of standard of baseline treatment for SLE from Day -1 or for any time during the study
* Active and clinically significant infection (bacterial, fungal, viral, or other) within 60 days prior to first dose of study drug. Clinically significant is defined as requiring systemic parenteral antibiotics or hospitalization
* A history of opportunistic infection, or a history of recurrent or severe disseminated herpes zoster or disseminated herpes simplex within the last 3 years
* Chronic viral hepatitis B (HBV) and hepatitis C (HCV), unless participant received curative treatment for HCV and has a documented negative viral load, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
* Cryptosporidium in the stool sample at screening
* White blood cells < 1,200/millimeters cubed (mm^3) (1.2 × 10^9/Liter [L]) at screening
* Absolute neutrophil count < 500/mm^3 at screening
* CD4+ count < 150/microliter (µL) at screening
* Platelets < 50,000/mm^3 (50 × 10^9/L) or < 35,000/mm^3 (35 × 10^9/L) if related to SLE, at screening
* Hemoglobin < 8 grams per deciliter (g/dL) or < 7 g/dL at screening if related to SLE
* Proteinuria > 3.0 g/day (3000 milligrams per day [mg/day]) at screening or equivalent level of proteinuria as assessed by protein/creatinine ratio (3 mg/mg or 339 milligrams per millimole [mg/mmol])
* Serum creatinine > 2.0 mg/dL at screening or creatinine clearance < 40 milliliters per minute (mL/minute) based on Cockcroft-Gault calculation
* Serum alanine aminotransferase and/or serum aspartate aminotransferase > 2 × the upper limit of normal (ULN) at screening, unless explicitly related to lupus based on the investigator's judgment
* Creatinine kinase > 3.0 × ULN at screening unless related to lupus myositis
* Total bilirubin > 1.5 × ULN at screening (unless related to Gilbert's syndrome)
* Any other laboratory test results that, in the opinion of the Investigator or the Sponsor or Sponsor's designee, might place a participant at unacceptable risk for participating in this study
* History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibodies (mAb) (eg, IgG protein) or molecules made of components of mAbs
* History substance and/or alcohol abuse, or dependence within the past 1 year, at the investigator's judgment
* History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer, or cervical cancer in situ resolved by excision)
* Any other severe acute or chronic medical or psychiatric condition, including recent (within the past year) medical conditions (eg, cardiovascular conditions, respiratory illnesses) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, Sponsor, or Sponsor's designee, would make the participant inappropriate for entry into this study
* Investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator, or participants who are employees of the sponsor or directly involved in the conduct of the trial
* Currently participating in, or who have participated in other interventional (drug or device) clinical study within 30 days or 5 half-lives of baseline, whichever is longer
* Recent (within the past 12 months) or active suicidal ideation or behavior based on participant responding "yes" to question 3, 4, or 5 on the Columbia Suicide severity Rating Scale
* Current or pending incarceration
* Current or pending compulsory detainment for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Currently taking a total daily dose of > 30 mg morphine or morphine equivalent
* Body mass index (BMI) ≥ 40.0

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (17):
  - Pinnacle Research Group, Anniston, Alabama
  - TriWest Research Associates, El Cajon, California
  - Valerius Medical Group and Research Center, Los Alamitos, California
  - Westlake Medical Research, Thousand Oaks, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Omega Research Consultants, DeBary, Florida
  - Centre for Rheumatology Immunology and Arthritis, Fort Lauderdale, Florida
  - Millennium Research, Ormond Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Clinic of Robert Hozman/Clinical Investigation Specialists, Inc., Skokie, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Aa Mrc Llc, Grand Blanc, Michigan
  - June DO PC, Lansing, Michigan
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Ramesh C. Gupta M.D., Memphis, Tennessee
  - Accurate Clinical Research Inc, Houston, Texas
- Argentina (4):
  - Hospital Militar Central - Servicio de Reumatología, Buenos Aires
  - Framingham Centro Medico, La Plata
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
  - Centro de Investigaciones Reumatologicas, San Miguel de Tucumán
- Bulgaria (3):
  - Diagnostic Consultative Center Sveti Georgi EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Medical Center - 1 - Sevlievo EOOD, Sevlievo
- Colombia (6):
  - Centro Integral de Reumatologia del Caribe CIRCARIBE S.A.S, Barranquilla
  - Preventive Care S.A.S., Bogotá
  - Medicity S.A.S., Bucaramanga
  - Servimed S.A.S., Bucaramanga
  - Clinica de Artritis Temprana, Cali
  - Hospital Pablo Tobon Uribe, Medellín
- Georgia (6):
  - V. Tsitlanadze Scientifically-Practical Rheumatology Center Ltd, Tbilisi
  - Research Institute of Clinical Medicine Ltd, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Mtskheta Street Clinic Ltd, Tbilisi
  - First Medical Center, Tbilisi
  - Multiprofile Clinic Consilium Medulla Ltd, Tbilisi
- Hungary (3):
  - Qualiclinic Kft., Budapest
  - DE Klinikai Központ, Debrecen
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Gyula
- Mexico (3):
  - Centro Integral en Reumatología S.A. de C.V. (CIRSA), Guadalajara
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - CLIDITER S.A. de C.V. (Centro de Investigación y Tratamiento de las Enfermedades Reumaticas), Mexico City
- Peru (5):
  - Hogar Clinica San Juan De Dios, Cayma
  - Centro de Investigación Clínica Trujillo E.I.R.L., La Libertad
  - Hospital Nacional Cayetano Heredia, Lima
  - Clinica San Juan Bautista, Lima
  - Instituto de Ginecología y Reproducción, Santiago de Surco
- Philippines (5):
  - Angeles University Foundation Medical Center, Angeles City
  - Southern Philippines Medical Center, Davao City
  - Mary Mediatrix Medical Center, Lipa City
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
- Poland (8):
  - Centrum Kliniczno - Badawcze J. Brzezicki, B. Gronkiewicz Brzezicka Spółka Lekarska, Elblag
  - Centrum Medyczne Plejady, Krakow
  - Centrum Nowoczesnych Terapii Dobry Lekarz sp. z o.o, Krakow
  - Centrum Medyczne AMED oddział w Łodzi, Lodz
  - NZOZ Lecznica MAK-MED, Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med Pawel Hrycaj, Poznan
  - SANUS Szpital Specjalistyczny sp. z o.o, Stalowa Wola
  - Reumatika-Centrum Reumatologii, Warsaw
- Romania (3):
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - Spitalul Clinic Judetean De Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic de Recuperare Iasi #2, Iași
- Ukraine (5):
  - National Scientific Center at Institute of Cardiology named after acad. M.D. Strazhesko, Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Odesa Regional Clinical Hospital, Odesa
  - Communal Non-Profit Enterprise "Ternopil University Clinic" of Ternopil Regional Council, Ternopil
  - Vinnytsia Regional Clinical Hospital, Vinnytsia

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in in the United States, Georgia, Bulgaria, Hungary, Poland, Argentina, Columbia, Mexico, Romania, Ukraine, Philippines and Peru. The first participant was screened on 10 January 2018 and last participant last visit occurred on 26, November 2020.
Groups:
- Phase 1b: Placebo: Participants were randomized to receive subcutaneous (SC) dose of placebo. Participants received a total of 7 SC monthly doses of placebo on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.
- Phase 1b: Cohort 1: BOS161721 20 mg: Participants were randomized to receive a 20 mg SC dose of BOS161721. Participants received a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
- Phase 1b: Cohort 2: BOS161721 60 mg: Participants were randomized to receive a 60 mg SC dose of BOS161721. Participants received a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270
- Phase 1b: Cohort 3: BOS161721 120 mg: Participants were randomized to receive a 120 mg SC dose of BOS161721. Participants received a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270
- Phase 2: Placebo: Participants were randomized to receive a SC dose of placebo (as determined from Phase 1b of the study). Participants received a total of 7 SC monthly doses of placebo on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
- Phase 2: BOS161721 120 mg: Participants were randomized to receive a 120 mg SC dose of BOS161721 (as determined from Phase 1b of the study). Participants received a total of 7 SC monthly doses of BOS161721 on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits on at Days 210, 240, and 270.
Period: Overall Study
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Started | 7 | 5 | 9 | 9 | 37 | 76
Completed | 5 | 5 | 8 | 9 | 30 | 71
Not Completed | 2 | 0 | 1 | 0 | 7 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 2 | 2
Not completed — Phase 1b: Pregnancy, Phase 2: fear of COVID-19 or local restrictions | 1 | 0 | 0 | 0 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Decision by Sponsor | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b: Placebo: Participants were randomized to receive a subcutaneous (SC) dose of placebo. Participants received a total of 7 SC monthly doses of placebo on Days 0, 30, 60, 90, 120, 150, and 180, followed by safety follow-up visits at Days 210, 240, and 270.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg | Phase 2: Placebo | Phase 2: BOS161721 120 mg | Total
Number analyzed (Participants) | 7 | 5 | 9 | 9 | 37 | 76 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In order to present the total data, the data for placebo (44 participants) and the data for BOS161721 (99 participants) have been presented in separate rows.
  years
    Placebo: number analyzed (Participants) | 7 | 0 | 0 | 0 | 37 | 0 | 44
    Placebo | 48.1 (17.67) |  |  |  | 45.7 (12.52) |  | 46.1 (13.25)
    BOS161721: number analyzed (Participants) | 0 | 5 | 9 | 9 | 0 | 76 | 99
    BOS161721 |  | 50.0 (8.51) | 49.3 (11.31) | 47.3 (10.43) |  | 44.5 (12.52) | 45.5 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 8 | 8 | 36 | 69 | 133
  Male | 0 | 0 | 1 | 1 | 1 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 17 | 32 | 53
  Not Hispanic or Latino | 6 | 4 | 7 | 9 | 20 | 44 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 3 | 6 | 7 | 18
  White | 5 | 5 | 9 | 6 | 20 | 45 | 90
  More than one race | 0 | 0 | 0 | 0 | 11 | 24 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Adverse Events (AEs)
Description: The safety, tolerability, and immunogenicity of repeat doses of BOS161721 (20, 60, and 120 mg) administered SC were assessed in adult participants with moderate to severe SLE on limited background standard of care treatment, in order to estimate the optimal dose.
Time Frame: Up to Day 270
Population: Safety Analysis Set (SS): Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least one evaluable post-baseline safety evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
Participants
  Any Treatment-Emergent Adverse Events (TEAE) | 4 | 2 | 7 | 8
  Related TEAE | 1 | 0 | 1 | 0
  Serious TEAE | 1 | 0 | 2 | 0
  Related Serious TEAE | 0 | 0 | 0 | 0
  Any Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or Higher TEAE | 4 | 2 | 6 | 7
  Any Related CTCAE Grade 2 or Higher TEAE | 1 | 0 | 0 | 0
  Any CTCAE Grade 3 TEAE | 1 | 1 | 2 | 0
  Any Related CTCAE Grade 3 or Higher TEAE | 0 | 0 | 0 | 0
  Any CTCAE Grade 4 TEAE | 0 | 0 | 0 | 0
  TEAE Leading to Discontinuation of Study Treatment | 0 | 0 | 0 | 0
  Related TEAE Leading to Discontinuation of Study Treatment | 0 | 0 | 0 | 0
  TEAE of Special Interest | 0 | 0 | 0 | 0
  Related TEAE of Special Interest | 0 | 0 | 0 | 0
  Dose-Limiting Toxicity | 0 | 0 | 0 | 0
  Related Dose-Limiting Toxicity | 0 | 0 | 0 | 0
  TEAE Resulting in Death | 0 | 0 | 0 | 0
  Related TEAE Resulting in Death | 0 | 0 | 0 | 0
  Injection Site Reaction | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: Number of Participants With an SLE Responder Index 4 (SRI-4) Response at Day 210
Description: The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLE Disease Activity Index 2000 (SLEDAI-2K), the British Isles Lupus Assessment Group (BILAG) 2004 Index and the Physician's Global Assessment (PGA). Response based on the SRI-4 is defined by: 1) ≥ 4-point reduction in the SLEDAI-2K total score; 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B) compared with baseline; and 3) no deterioration from baseline in the PGA by ≥ 30 millimeters. The SLEDAI-2K total score falls between 0 and 105, with higher scores representing increased disease activity.The SRI-4 response in participants with moderate to severe SLE is associated with broad improvements in clinical and participant-reported outcomes.
Time Frame: Day 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post-baseline efficacy evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants
  SRI-4 Response | 19 | 40
  ≥ 4-Point Reduction from Baseline in SLEDAI-2K Global Score | 19 | 40
  No New BILAG A or More than One BILAG B Organ Score Compared with Baseline | 27 | 68
  No Deterioration from Baseline in PGA by >=30mm | 27 | 68
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis: SRI-4 Response; Test type: Superiority; p = 0.8434, Pearson's chi-square test; Observed Difference vs. Placebo = 2.0, 90% CI 2-sided [-14.5 to 18.5]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis: >= 4-Point Reduction from Baseline in SLEDAI-2K Global Score; Test type: Superiority; p = 0.8434, Pearson's chi-square test; Observed Difference vs. Placebo = 2.0, 90% CI 2-sided [-14.5 to 18.5]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis: No New BILAG A or More than One BILAG B Organ Score Compared with Baseline; Test type: Superiority; p = 0.0141, Pearson's chi-square test; Observed Difference vs. Placebo = 17.7, 90% CI 2-sided [4.5 to 30.9]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis: No Deterioration from Baseline in PGA by >=30mm; Test type: Superiority; p = 0.0141, Pearson's chi-square test; Observed Difference vs. Placebo = 17.7, 90% CI 2-sided [4.5 to 30.9]

3. Secondary Outcome: Phase 1b: Maximum Observed Concentration (Cmax)
Description: The PK of BOS161721 was characterized and the optimal dose of BOS161721 was selected based on safety, tolerability, PK and PD data in participants with moderate to severe SLE.
Time Frame: Pre-dose: Days 0, 30, 60, 90, 120, 150, and 180. Post-dose: Days 0, 7, 15, 30, 180, 187, 195, 210, 240, and 270. Post-dose samples were collected at 4, 8, and 24 hours after study drug administration on Days 0, 30, and 180
Population: The PK population is defined as all participants who received at least 1 dose (partial or complete) of study treatment and had sufficient concentration data for the calculation of PK parameters. Here, number analyzed in each row signifies only the participants with available data for each dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 9 | 9
ng/mL
  Dose 1: number analyzed (Participants) | 4 | 8 | 9
  Dose 1 | 1160 (42.0) | 4610 (54.8) | 5500 (52.3)
  Dose 2: number analyzed (Participants) | 5 | 8 | 9
  Dose 2 | 1240 (23.9) | 5670 (35.7) | 7580 (45.1)
  Dose 7: number analyzed (Participants) | 5 | 8 | 9
  Dose 7 | 2580 (19.1) | 7820 (144) | 20300 (37.1)

4. Secondary Outcome: Phase 1b: First Time to Maximum Concentration (Tmax)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Day
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 9 | 9
Day
  Dose 1: number analyzed (Participants) | 4 | 8 | 9
  Dose 1 | 7.01 [6.99 to 12.00] | 7.00 [5.93 to 15.00] | 8.04 [6.95 to 17.04]
  Dose 2: number analyzed (Participants) | 5 | 8 | 9
  Dose 2 | 1.04 [1.00 to 29.02] | 1.00 [0.99 to 34.97] | 1.00 [1.00 to 33.03]
  Dose 7: number analyzed (Participants) | 5 | 8 | 9
  Dose 7 | 6.18 [5.03 to 20.04] | 3.55 [0.91 to 12.00] | 8.96 [1.00 to 28.06]

5. Secondary Outcome: Phase 1b: The Area Under the Plasma Concentration Versus Time Curve, From Time 0 to the Last Quantifiable Concentration (AUClast)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 9 | 9
day*ng/mL
  Dose 1: number analyzed (Participants) | 4 | 8 | 9
  Dose 1 | 25100 (40.4) | 89400 (51.7) | 124000 (40.5)
  Dose 2: number analyzed (Participants) | 5 | 8 | 9
  Dose 2 | 33600 (18.2) | 147000 (29.7) | 229000 (47.9)
  Dose 7: number analyzed (Participants) | 5 | 8 | 9
  Dose 7 | 155000 (17.9) | 460000 (173) | 1400000 (38.7)

6. Secondary Outcome: Phase 1b: Terminal Elimination Half-life (t1/2)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The PK population is defined as all participants who received at least 1 dose (partial or complete) of study treatment and had sufficient concentration data for the calculation of PK parameters. Here, overall number of participants analyzed signifies only the participants with available data for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 5 | 1
Day | 75.2 (19.9) | 66.3 (35.4) | 64.3 (NA) — Not calculated for 1 participant

7. Secondary Outcome: Phase 1b: Apparent Plasma Clearance After Extravascular Administration (CL/F)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/day
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 8 | 9
Liter/day | 0.289 (18.3) | 0.311 (179) | 0.218 (38.8)

8. Secondary Outcome: Phase 1b: Apparent Volume of Distribution After Extravascular Administration (Vz/F)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 5 | 5 | 1
Liter | 31.4 (33.2) | 18.5 (39.6) | 23.0 (NA) — Not calculated for 1 participant

9. Secondary Outcome: Phase 1b: Mean Change From Baseline in Phosphorylated Signal Transducer and Activator of Transcription 3 (pSTAT3)
Description: The optimal dose of BOS161721 was selected based on safety, tolerability, PK and pharmacodynamic (PD) data in participants with moderate to severe SLE.
Time Frame: Baseline (Day 0); Days 30, 44, 60, and 90 (pre-dose [trough] samples only)
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, number analyzed in each row signifies only the participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
Percentage
  % pSTAT3+ Lymphocytes - Stimulated, Day 30: number analyzed (Participants) | 6 | 5 | 8 | 9
  % pSTAT3+ Lymphocytes - Stimulated, Day 30 | 12.72 (25.172) | -41.80 (24.631) | -31.35 (20.281) | -25.73 (20.895)
  % pSTAT3+ Lymphocytes - Stimulated, Day 44: number analyzed (Participants) | 6 | 5 | 8 | 9
  % pSTAT3+ Lymphocytes - Stimulated, Day 44 | 18.45 (24.025) | -60.00 (19.672) | -32.99 (19.899) | -26.57 (20.856)
  % pSTAT3+ Lymphocytes - Stimulated, Day 60: number analyzed (Participants) | 6 | 5 | 8 | 9
  % pSTAT3+ Lymphocytes - Stimulated, Day 60 | -1.48 (19.129) | -59.46 (20.310) | -32.68 (19.214) | -25.91 (20.850)
  % pSTAT3+ Lymphocytes - Stimulated, Day 90: number analyzed (Participants) | 5 | 5 | 8 | 9
  % pSTAT3+ Lymphocytes - Stimulated, Day 90 | -15.94 (34.757) | -67.48 (15.630) | -33.03 (19.637) | -26.74 (20.962)

10. Secondary Outcome: Phase 1b: Mean Change From Baseline in Complement 3 (C3) and Complement (C4) Levels
Description: The optimal dose of BOS161721 was selected based on safety, tolerability, PK and PD data in participants with moderate to severe SLE.
Time Frame: Baseline (Day 0); Day 210
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram/Litre
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
gram/Litre
  C3, Day 210: number analyzed (Participants) | 5 | 5 | 8 | 9
  C3, Day 210 | 0.094 (0.2289) | -0.032 (0.0876) | 0.050 (0.3424) | -0.078 (0.2879)
  C4, Day 210: number analyzed (Participants) | 5 | 5 | 8 | 9
  C4, Day 210 | 0.024 (0.0391) | -0.038 (0.0370) | -0.007 (0.0783) | -0.024 (0.0410)

11. Secondary Outcome: Phase 1b: Mean Change From Baseline in Leukocyte Immunophenotype
Description: as for outcome 10
Time Frame: Baseline (Day 0); Day 180
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Change in percentage of cells
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
Change in percentage of cells
  CD19+% of CD45+ Lymphocytes | -2.07 (3.201) | -5.34 (4.663) | -0.39 (4.201) | 0.27 (3.481)
  CD25+CD127-% of CD4+CD8- | -1.03 (1.388) | -0.22 (2.406) | -0.38 (1.495) | -1.08 (2.266)
  CD4+CD8-% of CD3+ | -1.01 (10.866) | -3.08 (5.272) | 0.88 (7.434) | -5.04 (7.671)
  CD56+% OF CD45+ Lymphocytes | -0.56 (2.093) | -5.76 (4.231) | -2.38 (2.461) | 2.04 (7.984)
  CD8+CD4-% of CD3+ | -3.00 (7.792) | -1.38 (4.467) | -2.92 (5.010) | -0.24 (6.517)
  CXCR5+% of CD25+CD127- | 0.20 (4.676) | 7.02 (3.371) | 10.62 (11.963) | 0.63 (5.915)
  CXCR5+% of CD4+CD8- | 0.81 (12.373) | 15.18 (7.564) | 13.14 (16.091) | -0.69 (7.208)
  ICOS+% of CD25+CD127- | 8.59 (10.618) | 1.56 (3.840) | 12.93 (11.905) | 4.27 (17.059)
  ICOS+% of CD4+CD8- | 3.93 (6.906) | 0.14 (5.227) | 5.01 (5.053) | 0.54 (15.534)
  IgD+C27-% of CD19+ | 0.20 (7.127) | 2.42 (5.882) | -1.07 (4.748) | -0.80 (6.031)
  IgD+CD27+% of CD19+ | 1.29 (1.785) | -3.24 (6.080) | -1.24 (2.823) | 1.00 (3.260)
  IgD+CD27-CD38++CD24++% of CD19+ | 0.50 (1.262) | 0.56 (1.688) | -0.42 (2.351) | 0.16 (1.385)
  IgD-CD27+% of CD19+ | -0.21 (3.866) | -0.48 (3.891) | 2.02 (3.751) | 0.70 (3.740)
  IgD-CD27+CD38++CD138+% of CD19+ | 0.03 (0.049) | 0.04 (0.089) | 0.08 (0.172) | -0.02 (0.130)
  IgD-CD27+CD38++CD138-% of CD19+ | -0.20 (0.432) | -0.20 (0.354) | 0.59 (1.437) | -0.63 (1.081)
  IgD-CD27-% of CD19+ | -1.29 (2.963) | 1.36 (2.373) | 0.32 (2.059) | -0.83 (1.648)
  PD-1+% of CD25+CD127- | 0.31 (6.093) | 3.30 (5.039) | 7.41 (6.064) | -8.49 (13.258)
  PD-1+% of CD4+CD8- | -0.07 (6.366) | 4.14 (4.146) | 6.39 (5.882) | -9.01 (13.036)

12. Secondary Outcome: Phase 1b: Mean Change From Baseline in Anti-double-stranded DNA (dsDNA) Autoantibodies at Each Visit
Description: as for outcome 10
Time Frame: Baseline (Day 0); Days 30, 60, 90, 120, 150, 180, 210, 240, and 270
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International units per millilitre
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
International units per millilitre
  Day 30: number analyzed (Participants) | 7 | 5 | 8 | 9
  Day 30 | -1.11 (3.504) | 0.48 (0.410) | 5.34 (9.053) | -11.51 (32.444)
  Day 60: number analyzed (Participants) | 7 | 5 | 8 | 9
  Day 60 | -1.81 (5.048) | 0.40 (0.376) | 8.06 (18.430) | -6.11 (15.612)
  Day 90: number analyzed (Participants) | 6 | 5 | 8 | 9
  Day 90 | 0.15 (0.448) | 0.00 (0.187) | 19.31 (48.594) | -13.44 (35.152)
  Day 120: number analyzed (Participants) | 6 | 5 | 8 | 9
  Day 120 | -0.02 (0.270) | 0.41 (0.598) | 12.30 (35.583) | -15.58 (47.248)
  Day 150: number analyzed (Participants) | 5 | 5 | 8 | 9
  Day 150 | -0.03 (0.199) | 0.62 (0.709) | 17.39 (50.086) | -11.18 (38.152)
  Day 180 | -2.13 (5.905) | 0.52 (0.584) | 8.00 (21.169) | -17.13 (49.897)
  Day 210: number analyzed (Participants) | 5 | 5 | 8 | 9
  Day 210 | 0.05 (0.359) | 0.07 (0.540) | 6.76 (20.173) | -17.96 (50.274)
  Day 240: number analyzed (Participants) | 5 | 5 | 8 | 9
  Day 240 | 0.07 (0.428) | 0.34 (1.117) | 6.81 (21.903) | -18.35 (47.898)
  Day 270: number analyzed (Participants) | 7 | 5 | 8 | 9
  Day 270 | -1.94 (4.974) | 0.37 (0.700) | 7.99 (24.116) | -9.71 (27.833)

13. Secondary Outcome: Phase 1b: Mean Change From Baseline in Anti-Sjögren's Syndrome A and B (SSA, SSB)
Description: The optimal dose of BOS161721 was selected based on safety, tolerability, PK and PD data in subjects with moderate to severe SLE.
Time Frame: Baseline (Day 0); Day 180
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and have at least 1 evaluable post baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
U/mL
  La Antibody | 0.04 (0.175) | 0.11 (0.108) | 1.02 (2.639) | 0.47 (1.668)
  Sjogrens SS-A52 Antibody | -0.04 (0.128) | 0.05 (0.112) | 0.19 (0.567) | -2.25 (4.861)
  Sjogrens SS-A60 Antibody | 0.00 (0.000) | 0.00 (0.000) | -2.62 (7.867) | -4.36 (8.684)

14. Secondary Outcome: Phase 1b: Mean Change From Baseline in Anti-Smith Antibody (Sm)
Description: as for outcome 13
Time Frame: Baseline (Day 0); Day 180
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
U/mL | -1.87 (4.827) | 0.74 (0.391) | -3.21 (9.419) | 3.61 (19.504)

15. Secondary Outcome: Phase 1b: Mean Change From Baseline in Antiphospholipid (APL) Autoantibodies (Beta 2 Glycoprotein, Cardiolipin IgG)
Description: as for outcome 10
Time Frame: Baseline (Day 0); Day 180
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 7 | 5 | 9 | 9
U/mL
  Anti-Cardiolipin IgG Antibody | -0.03 (0.412) | 3.55 (5.559) | 0.07 (0.585) | -0.42 (0.180)
  Beta-2 Glycoprotein 1 IgG Antibody | -0.11 (0.358) | -7.48 (23.684) | -0.14 (0.882) | 0.02 (0.787)

16. Secondary Outcome: Phase 1b: Mean Change From Baseline in Abrogation of IL-21 Gene Signature
Description: as for outcome 10
Time Frame: Baseline (Day 0); Days 15, 90, 180, and 270
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and have at least 1 evaluable post baseline efficacy evaluation. Data were not collected for this outcome measure.
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Phase 2: Number of Participants With an SRI-4, SRI-5, and SRI-6 Response at Each Visit
Description: The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from the SLE Disease Activity Index 2000 (SLEDAI-2K) and the British Isles Lupus Assessment Group (BILAG) 2004 Index. Response based on the SRI-4 is defined by: 1) ≥ 4-point reduction in the SLEDAI-2K global score; 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B); and 3) no deterioration from baseline in the Physician's Global Assessment (PGA) by ≥ 30 millimeters. The SRI-4 response in participants with moderate to severe SLE is associated with broad improvements in clinical and participant-reported outcomes. SRI-5 and SRI-6 are composite indices of SLE disease improvement that consist of scores derived from the SLEDAI-2K and the BILAG 2004 Index. The SRI-5 and SRI-6 are computed with a minimal five-point or six-point improvement in SLEDAI-2K being required, respectively.
Time Frame: Days 30, 60, 90, 120, 150, 180, 210, 240, and 270
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants
  SRI-4, Day 30: number analyzed (Participants) | 36 | 73
  SRI-4, Day 30 | 5 | 0
  SRI-4, Day 60: number analyzed (Participants) | 35 | 71
  SRI-4, Day 60 | 11 | 15
  SRI-4, Day 90: number analyzed (Participants) | 35 | 65
  SRI-4, Day 90 | 15 | 24
  SRI-4, Day 120: number analyzed (Participants) | 35 | 66
  SRI-4, Day 120 | 17 | 29
  SRI-4, Day 150: number analyzed (Participants) | 35 | 71
  SRI-4, Day 150 | 19 | 35
  SRI-4, Day 180: number analyzed (Participants) | 35 | 72
  SRI-4, Day 180 | 20 | 37
  SRI-4, Day 210 | 19 | 40
  SRI-5, Day 30: number analyzed (Participants) | 36 | 73
  SRI-5, Day 30 | 2 | 0
  SRI-5, Day 60: number analyzed (Participants) | 35 | 71
  SRI-5, Day 60 | 1 | 10
  SRI-5, Day 90: number analyzed (Participants) | 35 | 65
  SRI-5, Day 90 | 3 | 15
  SRI-5, Day 120: number analyzed (Participants) | 35 | 66
  SRI-5, Day 120 | 8 | 15
  SRI-5, Day 150: number analyzed (Participants) | 35 | 71
  SRI-5, Day 150 | 15 | 22
  SRI-5, Day 180: number analyzed (Participants) | 35 | 72
  SRI-5, Day 180 | 14 | 29
  SRI-5, Day 210 | 17 | 29
  SRI-6, Day 30: number analyzed (Participants) | 36 | 73
  SRI-6, Day 30 | 1 | 0
  SRI-6, Day 60: number analyzed (Participants) | 35 | 71
  SRI-6, Day 60 | 1 | 10
  SRI-6, Day 90: number analyzed (Participants) | 35 | 65
  SRI-6, Day 90 | 3 | 15
  SRI-6, Day 120: number analyzed (Participants) | 35 | 66
  SRI-6, Day 120 | 8 | 14
  SRI-6, Day 150: number analyzed (Participants) | 35 | 71
  SRI-6, Day 150 | 15 | 22
  SRI-6, Day 180: number analyzed (Participants) | 35 | 72
  SRI-6, Day 180 | 14 | 28
  SRI-6, Day 210 | 17 | 29

18. Secondary Outcome: Phase 2: Number of Participants With a Sustained Reduction From Baseline of Oral Corticosteroid (CS) (≤ 7.5 mg/Day and < Day 0 Dose) Between Day 150 and Day 210
Description: Effect of BOS161721 compared with placebo for response on clinical indicators of SLE activity was assessed in adult participants with moderate to severe SLE on limited background standard of care treatment.
Time Frame: Day 150 to Day 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, overall number of participants analyzed signifies only the number of participants taking oral corticosteroids at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 25 | 67
Participants | 7 | 17
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.7985, Pearson's chi-square test; Observed Difference vs. Placebo = -2.6, 90% CI 2-sided [-19.8 to 14.5]

19. Secondary Outcome: Phase 2: Number of Participants With New or Recurrent BILAG Flares (≥ 1 Qualifying BILAG A or > 1 Qualifying BILAG B) Through Day 210
Description: The BILAG-2004 index is an organ-specific 97-question assessment based on the principle of the doctor's intent to treat. Only clinical features attributable to SLE disease activity were recorded and based on the participant's condition in the last 4 weeks compared with the previous 4 weeks. It was scored as not present (0), improved (1), the same (2), worse (3), or new (4). Disease activity was graded separately for 9 body systems to 5 different grades (A to E) as follows: A is very active disease, B is moderate activity, C is mild stable disease, D is inactive now but previously active, and E indicates the organ was never involved. A shift from BILAG-2004 Grade A or B to a lower grade indicates a clinically relevant change in disease activity as the BILAG-2004 grades mirror the decision points for treatment interventions.
Time Frame: Days 30, 60, 90, 120, 150, 180, 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, number analyzed in each row signifies only the number of participants with a post-baseline BILAG assessment at any time (overall assessment) or at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants
  Overall | 6 | 7
  Day 30: number analyzed (Participants) | 36 | 73
  Day 30 | 1 | 2
  Day 60: number analyzed (Participants) | 33 | 66
  Day 60 | 0 | 0
  Day 90: number analyzed (Participants) | 33 | 65
  Day 90 | 2 | 0
  Day 120: number analyzed (Participants) | 31 | 65
  Day 120 | 1 | 0
  Day 150: number analyzed (Participants) | 32 | 71
  Day 150 | 0 | 1
  Day 180: number analyzed (Participants) | 34 | 71
  Day 180 | 1 | 3
  Day 210: number analyzed (Participants) | 31 | 72
  Day 210 | 0 | 1
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Overall; Test type: Superiority; p = 0.3498, Pearson's chi-square test; Observed Difference vs. Placebo = -6.9, 90% CI 2-sided [-22.9 to 9.8]

20. Secondary Outcome: Phase 2: Number of Participants With Physician's Global Assessment (PGA) Worsening
Description: The PGA is used to assess Investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". PGA worsening is defined as an increase of ≥ 30 mm from baseline.
Time Frame: Days 30, 60, 90, 120, 150, 180, and 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, number analyzed in each row signifies the number of participants with a post-baseline PGA assessment at any time (overall assessment) or at the given timepoint (by visit assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants
  Overall | 13 | 10
  Day 210 | 10 | 7
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical analysis for Overall; Test type: Superiority; p = 0.0072, Pearson's chi-square test; Observed Difference vs. Placebo = -21.8, 90% CI 2-sided [-36.2 to -7.4]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Day 210; Test type: Superiority; p = 0.0141, Pearson's chi-square test; Observed Difference vs. Placebo = -17.7, 90% CI 2-sided [-30.9 to -4.5]

21. Secondary Outcome: Phase 2: Number of Participants With a BILAG-based Composite Lupus Assessment (BICLA) Response at Day 210
Description: The BICLA is a responder index developed to measure response to therapy, and it includes scores from the BILAG, SLEDAI-2K, and Physician's Global Assessment (PGA). BICLA response is defined as: 1) at least 1 gradation of improvement in baseline BILAG 2004 scores in all body systems with moderate disease activity at entry (eg, all B [moderate disease] scores falling to C [mild], or D [no activity]); 2) no new BILAG A or more than 1 new BILAG B scores; 3) no worsening of total SLEDAI-2K score from baseline; 4) ≤ 10% deterioration in PGA score; and 5) no treatment failure. The PGA is measured on a 0 to 100 mm scale with score 0 to be No Disease Activity and score 100 to be the most Severe Disease Activity.
Time Frame: Day 210
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants | 12 | 28
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.6107, Pearson's chi-square test; Observed Difference vs. Placebo = 4.9, 90% CI 2-sided [-10.7 to 20.5]

22. Secondary Outcome: Phase 2: Number of Participants With a Cutaneous Lupus Erythematosus Area and Severity Index (CLASI) Response at Day 210
Description: The CLASI is a comprehensive tool for assessment of disease activity (CLASI-A) in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. Response is defined as at least 50% improvement from baseline in "A" scores. This assessment was applied to all participants as all were required to have cutaneous disease activity. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
Time Frame: Day 210
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants | 16 | 44
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.1237, Pearson's chi-square test; Observed Difference vs. Placebo = 15.4, 90% CI 2-sided [-0.9 to 31.8]

23. Secondary Outcome: Phase 2: Number of Participants With Medication Failures
Description: as for outcome 18
Time Frame: Days 30, 60, 90, 120, 150, 180, and 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, number analyzed in each row signifies the number of participants evaluable at any time (overall assessment) or at the given timepoint (by visit assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Participants
  Overall | 9 | 8
  Day 210: number analyzed (Participants) | 33 | 72
  Day 210 | 7 | 5
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Overall; Test type: Superiority; p = 0.0581, Pearson's chi-square test; Observed Difference vs. Placebo = -13.7, 90% CI 2-sided [-26.7 to -0.7]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Day 210; Test type: Superiority; p = 0.0471, Pearson's chi-square test; Observed Difference vs. Placebo = -14.3, 90% CI 2-sided [-31.2 to 3.2]

24. Secondary Outcome: Phase 2: Mean Change From Baseline in CLASI at Day 210
Description: The CLASI is a comprehensive tool for the assessment of disease activity (CLASI-A) and damage (CLASI-B) in cutaneous lupus, shown to be valid, reliable, and sensitive to changes in disease activity. Response is defined as 50% improvement from baseline in "A" or "B" scores. This assessment was applied to all participants as all were required to have cutaneous disease activity. The total score represents the sum of the individual scores and ranges from 0 to 70 (CLASI-A) and 0 to 58 (CLASI-B). Higher scores are awarded for more severe manifestations. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline, Day 210
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
score on a scale
  CLASI-A (Total Activity) | -4.8 (4.08) | -5.2 (4.62)
  CLASI-B (Total Damage) | -0.6 (2.61) | -0.2 (0.90)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for CLASI-A (Total Activity); Test type: Superiority; p = 0.6596, ANCOVA; Treatment Difference (BOS161721-Placebo) = -0.3, 90% CI 2-sided [-1.63 to 0.94], Standard Error of Mean 0.78 — This is based on LS Means
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for CLASI-B (Total Damage); Test type: Superiority; p = 0.4105, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.3, 90% CI 2-sided [-0.27 to 0.81], Standard Error of Mean 0.33 — This is based on LS Means

25. Secondary Outcome: Phase 2: Mean Change From Baseline in PGA
Description: The PGA is used to assess Investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients".
Time Frame: Baseline, Day 210
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
score on a scale | -29.2 (20.69) | -28.7 (20.35)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Day 210; Test type: Superiority; p = 0.8546, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.8, 90% CI 2-sided [-6.07 to 7.58], Standard Error of Mean 4.11 — This is based on LS Means

26. Secondary Outcome: Phase 2: Mean Change From Baseline in the Total Number of Swollen Joints, Tender Joints, and Active Joints (Swelling and Tenderness in the Same Joint) in the American College of Rheumatology-28 (ACR-28) Joint Count
Description: The ACR-28 joint count evaluated the number of tender and swollen joints in the shoulder, elbow, wrist, hand, and knee joints. Joints of the feet were excluded. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline, Day 210
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Number of swollen/tender/active joints
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Number of swollen/tender/active joints
  Sum of Swelling | -6.8 (5.17) | -5.9 (5.05)
  Sum of Tenderness | -8.3 (7.00) | -7.2 (5.57)
  Sum of Active Joints | -6.5 (5.54) | -5.6 (4.65)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Sum of Swelling for Day 210; Test type: Superiority; p = 0.4455, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.5, 90% CI 2-sided [-0.63 to 1.71], Standard Error of Mean 0.70 — This is based on LS Means
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Sum of Tenderness for Day 210; Test type: Superiority; p = 0.3367, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.9, 90% CI 2-sided [-0.65 to 2.47], Standard Error of Mean 0.94 — This is based on LS Means
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Sum of Active Joints for Day 210; Test type: Superiority; p = 0.2550, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.8, 90% CI 2-sided [-0.34 to 1.86], Standard Error of Mean 0.66 — This is based on LS Means

27. Secondary Outcome: Phase 2: Mean Change From Baseline in SLEDAI-2K at Day 210
Description: The SLEDAI-2K is a validated instrument that measures disease activity in SLE participants at the time of the visit and in the previous 30 days. It is a global index and includes 24 clinical and laboratory variables that are weighted by the type of manifestation, but not by severity. The total score falls between 0 and 105, with higher scores representing increased disease activity. A SLEDAI -2K of 6 or more generally represents moderately to severely active disease.
  Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline, Day 210
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
score on a scale | -4.7 (3.71) | -3.9 (3.31)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.2498, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.8, 90% CI 2-sided [-0.34 to 1.93], Standard Error of Mean 0.68 — This is based on LS Means

28. Secondary Outcome: Phase 2: Mean Change From Baseline in Systemic Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index
Description: The SLICC/ACR damage index is a validated instrument to assess damage, defined as irreversible impairment, continuously persistent for 6 months (ascertained by clinical assessment), occurring since the onset of lupus, and it is based on a weighted scoring system. This index records damage occurring in participants with SLE regardless of cause, with demonstrated content, face, criterion, and discriminant validity. A score of 0=no damage. Total maximum score is 47 and increasing score indicates increasing disease severity.
Time Frame: Baseline; Day 180
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Here, overall number of participants analyzed signifies only the participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 30 | 67
score on a scale | 0 (0) | 0.1 (0.24)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Statistical Analysis for Day 180; Test type: Superiority; p = 0.2558, ANCOVA; Treatment Difference (BOS161721-Placebo) = 0.0, 90% CI 2-sided [-0.02 to 0.12], Standard Error of Mean 0.04 — This is based on LS Means

29. Secondary Outcome: Phase 2: Time to Medication Failure
Description: Participants who received prohibited medications or undergo unallowable corticosteroid (CS) usage were considered "medication failures".
Time Frame: Up to Day 270
Population: as for outcome 11
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Days | NA [NA to NA] — Median was not established based on the number of medication failures observed. | NA [NA to NA] — Median was not established based on the number of medication failures observed.
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.0479, Log Rank; Hazard Ratio (HR) = 0.39, 90% CI 2-sided [0.18 to 0.88] — Hazard rate of BOS161721 120 mg / Hazard rate of placebo

30. Secondary Outcome: Mean Percent Change in CS Administration From the Baseline Day 0 Dose Through Day 210 in Participants Receiving ≥ 7.5 mg/Day Prednisone Equivalent at Day 0
Description: The percent reduction in CS administration from Day 0 through Day 210 was determined based on the average daily CS usage.
Time Frame: Baseline; Day 210
Population: Full Analysis Set: Defined as all participants who received at least 1 dose (partial or complete) of study treatment and had at least 1 evaluable post baseline efficacy evaluation. Participants in the Full Analysis Set who received >= 7.5 mg/day prednisone equivalent at Day 0 were included. Here, overall number of participants analyzed signifies only the participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Reduction in Dose (mg/day)
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 13 | 45
Percent Reduction in Dose (mg/day) | -36.61 (22.389) | -21.49 (26.950)

31. Secondary Outcome: Phase 2: Duration of Longest SRI-4 Response
Description: The SRI-4 is a composite index of SLE disease improvement that consists of scores derived from SLEDAI-2K, BILAG 2004 Index and PGA. Response based on the SRI-4 is defined by: 1) ≥ 4-point reduction in the SLEDAI-2K total score; 2) no new severe disease activity (BILAG A organ score) or more than 1 new moderate organ score (BILAG B) compare with baseline; and 3) no deterioration from baseline in the PGA by ≥ 30 millimeters. The total SLEDAI-2K score falls between 0 and 105, with higher scores representing increased disease activity. The PGA is used to assess Investigator's general impression on the patient's overall status of SLE disease activity via visual analogue scale (100 mm) with 0 being "very good, asymptomatic and no limitation of normal activities" with 100 mm being "most severe possible disease ever seen in all SLE patients". The SRI-4 response in participants with moderate to severe SLE is associated with broad improvements in clinical and participant-reported outcomes.
Time Frame: Up to Day 270
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Days | 119.8 (68.26) | 124.2 (68.48)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.7898, ANOVA; Treatment Difference (BOS161721-Placebo) = 4.4, 90% CI 2-sided [-22.92 to 31.70], Standard Error of Mean 16.40 — This is based on LS Means

32. Secondary Outcome: Phase 2: Time to First BILAG Flare (≥ 1 New or Recurrent BILAG A or > 1 New or Recurrent BILAG B) Relative to Baseline Through Day 210
Description: as for outcome 19
Time Frame: Baseline; Day 210
Population: as for outcome 11
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 75
Days | NA [NA to NA] — Median was not established based on the number of BILAG flares observed. | NA [NA to NA] — Median was not established based on the number of BILAG flares observed.
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: BOS161721 120 mg; Test type: Superiority; p = 0.0083, Log-Rank Test (2-Sided); Hazard Ratio (HR) = 0.33, 90% CI 2-sided [0.16 to 0.68] — Hazard rate of BOS161721 120mg / Hazard rate of placebo

33. Secondary Outcome: Phase 2: Number of Participants With AEs
Description: The safety and tolerability of repeat doses of BOS161721 (120 mg) administered SC were assessed in adult participants with moderate to severe SLE on limited background standard of care treatment.
Time Frame: Up to Day 270
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: BOS161721 120 mg
Number analyzed (Participants) | 37 | 76
Participants
  Any TEAE | 23 | 44
  Related TEAE | 4 | 8
  Serious TEAE | 3 | 2
  Related Serious TEAE | 0 | 0
  Any CTCAE Grade 2 or Higher TEAE | 16 | 25
  Any Related CTCAE Grade 2 or Higher TEAE | 0 | 3
  Any CTCAE Grade 3 TEAE | 3 | 6
  Any Related CTCAE Grade 3 or Higher TEAE | 0 | 0
  Any CTCAE Grade 4 TEAE | 0 | 0
  Any Related CTCAE Grade 4 TEAE | 0 | 0
  TEAE Leading to Discontinuation of Study Treatment | 1 | 0
  Related TEAE Leading to Discontinuation of Study Treatment | 0 | 0
  TEAE of Special Interest | 0 | 1
  Related TEAE of Special Interest | 0 | 0
  Dose-Limiting Toxicity | 0 | 0
  Related Dose-Limiting Toxicity | 0 | 0
  TEAE Resulting in Death | 0 | 0
  Related TEAE Resulting in Death | 0 | 0
  Injection Site Reaction | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to Day 270
Arm/Group | Phase 1b: Placebo | Phase 1b: Cohort 1: BOS161721 20 mg | Phase 1b: Cohort 2: BOS161721 60 mg | Phase 1b: Cohort 3: BOS161721 120 mg | Phase 2: Placebo | Phase 2: BOS161721 120 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/9 | 0/9 | 0/37 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/5 | 2/9 | 0/9 | 3/37 | 2/76
Other Adverse Events (participants affected / at risk) | 4/7 | 2/5 | 7/9 | 8/9 | 22/37 | 44/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Placebo (N=7) | Phase 1b: Cohort 1: BOS161721 20 mg (N=5) | Phase 1b: Cohort 2: BOS161721 60 mg (N=9) | Phase 1b: Cohort 3: BOS161721 120 mg (N=9) | Phase 2: Placebo (N=37) | Phase 2: BOS161721 120 mg (N=76)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exomphalos (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Placebo (N=7) | Phase 1b: Cohort 1: BOS161721 20 mg (N=5) | Phase 1b: Cohort 2: BOS161721 60 mg (N=9) | Phase 1b: Cohort 3: BOS161721 120 mg (N=9) | Phase 2: Placebo (N=37) | Phase 2: BOS161721 120 mg (N=76)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 7 (9)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 4 (4) | 4 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected Bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media Acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (5)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sjogren's Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (6)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Adnexa Uteri Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03371251/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03371251/SAP_001.pdf